CLINICAL TRIAL: NCT06516302
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase III Clinical Trial Evaluating the Efficacy, Safety, and Immunogenicity of GR1802 in Participants With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: A Study of GR1802 in Participants With Chronic Sinusitis With Nasal Polyps
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1802-007
Record Dates: First submitted 2024-07-08; First posted 2024-07-23 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GR1802 group (Experimental): GR1802 300mg is administrated every 2 weeks (first dose doubled) for a total of 26 doses, of which an additional 2 ml of placebo is given at week 24.
  Interventions: Drug: GR1802
- placebo group (Placebo Comparator): Placebo is administered every 2 weeks for the first 16 weeks. GR1802 is given every 2 weeks from week 24 to W50.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GR1802 — GR1802 will be administered SC.
  Arms: GR1802 group
Drug: Placebo — The placebo will be administered SC.
  Arms: placebo group

SUMMARY:
The goal of this clinical trial is to learn if GR1802 works to treat severe chronic rhinosinusitis with nasal polyps (CRSwNP) in adults. It will also learn about the safety of GR1802. The main questions it aims to answer are:

1. Does GR1802 reduce the need for surgery and systemic corticosteroid use？
2. What medical problems do participants have when taking GR1802?

Researchers will compare GR1802 to a placebo (a look-alike substance that contains no drug) to see if GR1802 works to treat CRSwNP.

Participants will:

Take GR1802 or a placebo once every 2 weeks for 13months. Visit the clinic once every 2 weeks for checkups and tests. Keep a diary of their symptoms and the dosage and number of times they use mometasone furoate nasal spray.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, multi-center clinical trial was designed. The clinical trial was divided into 4 stages: screening/introduction period, double-blind treatment period , maintenance treatment period and safety follow-up period.

The clinical trial aimed to evaluate the efficacy, safety and immunogenicity of GR1802 injection in CRSwNP participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as CRSwNP and treated with systemic glucocorticoid within 2 years before screening; and/or those who had undergone surgery for nasal polyps before screening.
* An endoscopic bilateral NPS at screening/lead-in period and the baseline period of at least 5 out of a maximum score of 8 (with a minimum socre of 2 in each nasal cavity).
* Nasal congestion/blockade/obstruction with moderate or severe symptom severity at at screening period (score 2 or 3 ) .
* Willing to sign an informed consent, able to comply with clinic visits and study-related procedures as per protocol.

Exclusion Criteria:

* Biologic therapy within 5 half-lives or within 10 weeks before baseline.
* Anti-IL-4Rα antibody before screening.
* An experimental drug within 5 half-lives or 1 months before baseline.
* Systemic immunosuppressant to treat inflammatory disease or autoimmune disease within 2 months or 5 half-lives before baseline.
* Initiation of allergen immunotherapy within 3 months before screening.
* Participants receiving leukotriene antagonist/modifier before screening unless on continous treatment for at least 30 days.
* Participants with FEV1 50% or less of predicted normal were excluded.
* Participants who have undergone any intranasal and/or sinus surgery within 6 months before screening.
* Acute sinusitis or upper respiratory infection within a defined time period before screening.
* A nasal cavity tumor (malignant or benign).
* Evidence of fungal rhinosinusitis.
* Presence of another diagnosis associated with nasal polyps (i.e., eosinophilic granulomatosis with polyangiitis, granulomatosis with polyangiitis, Young's syndrome, cystic fibrosis).
* Rhinitis medicamentosa.
* Nasal septal deviation occluding at least one nostril.
* Antrochoanal polyps.
* Pregnant or lactating woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in nasal polyps score at week 24. | At week 24
  Nasal polyps score score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Change from baseline in nasal congestion score at week 24. | At week 24
  Nasal congestion score (0-3), higher score means worse nasal symptom.

SECONDARY OUTCOMES:
Change from baseline in reduction/loss of smell at weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56 and 60. | From baseline to week 60
  The reduction/loss of smell severity was reported by the participant on a daily basis using a 0 to 3 categorical scale. Higher score means a worse sense of smell.
Change from baseline in nasal discharge (anterior/posterior) at weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56 and 60. | From baseline to week 60
  The nasal discharge severity was reported by the participant on a daily basis using a 0 to 3 categorical scale. Higher score means a worse nasal symptom.
Change from baseline in Total Nasal Symptom Score (TNSS) at weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56 and 60. | From baseline to week 60
  TNSS score (0-9). Higher score means worse nasal symptom.
Change from baseline in nasal endoscopy nasal polyps score in participants with a high power field of vision < 55 eosinophil granulocytes in nasal polyp tissue at week 24. | At week 24
  Nasal polyps score score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Change from baseline in nasal congestion score in participants with a high power field of vision < 55 eosinophil granulocytes in nasal polyp tissue at week 24. | At week 24
  Nasal congestion score (0-3), higher score means worse nasal symptom.
Change from baseline in nasal polyps score at weeks 2、4、8、16、32、40、52 and 60. | From baseline to week 60
  Nasal polyps score score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Proportion of participants with improvement by at least 1 point in nasal polyps score at weeks 2、4、8、16、24、32、40、52 and 60. | From baseline to week 60
  Nasal polyps score score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Proportion of participants with improvement by at least 2 point in nasal polyps score at weeks 2、4、8、16、24、32、40、52 and 60. | From baseline to week 60
  Nasal polyps score score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Time to first response (≥1 point improvement) in nasal polyps score. | From baseline to week 60
  Nasal polyps score score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Change from baseline in nasal congestion score at weeks 4、8、12、16、20、28、32、36、40、44、48、52、56 and 60. | From baseline to week 60
  Nasal congestion score (0-3), higher score means worse nasal symptom.
Proportion of participants with improvement by at least 1 point in nasal congestion score at weeks 4、8、12、16、20、24、28、32、36、40、44、48、52、56 and 60. | From baseline to week 60
  Nasal congestion score (0-3), higher score means worse nasal symptom.
Proportion of participants with improvement by at least 2 point in nasal congestion score at weeks 4、8、12、16、20、24、28、32、36、40、44、48、52、56 and 60. | From baseline to week 60
  Nasal congestion score (0-3), higher score means worse nasal symptom.
Change from baseline in Lund-Mackay score at week 24 and 52. | From baseline to week 60
  The range of LM score is 0-24. Higher score means worse rhinosinusitis.
Change from baseline in 22-item Sinonasal Outcome Test (SNOT-22) at weeks 2, 4, 8, 16, 24, 32, 40, 52 and 60. | From baseline to week 60
  The range of SNOT-22 score is 0 to 110. Higher scores indicating more severe disease.
Change from baseline in University of Pennsylvania Smell Identification Test (UPSIT) at weeks 2, 4, 16, 24, 32, 40, 52 and 60. | From baseline to week 60
  UPSIT score (0-40). Higher score means better sense of smell.
Change from baseline in five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) at weeks 4、16、24、40、52 and 60. | From baseline to week 60
  The EQ-5D-5L descriptive system comprises five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), and each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the five dimensions.
Safety parameters. | From baseline to week 60
  Incidence of treatment-emergent adverse events (TEAEs), incidence of treatment-emergent serious AEs (TESAEs), etc.
Pharmacokinetics, include Ctrough, etc. | From baseline to week 60
  GR1802 concentrations were measured in CRSwNP population using sparse sampling (samples collected at predose, during treatment, and the follow up period).
Pharmacodynamics. | From baseline to week 60
  Levels of the type 2 inflammation biomarkers were assessed as markers for disease activity/severity.
Immunogenicity, include ADA and Nab. | From baseline to week 60
  Anti GR1802 antibody status was determined at baseline and at prespecified time points.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Doctor, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No